CLINICAL TRIAL: NCT06013761
Title: Monocentric Randomized Experimental Pilot Trial Investigating the Influence of Intermittent Fasting According to the 16:8 Method With and Without Medium-chain Triglycerides (MCTs) on Seizure Frequency, Biomarkers and Neural Networks in Patients With Drug-resistant Epilepsy
Brief Title: IF-MCT 16:8: Investigating the Influence of Intermittent Fasting With and Without MCTs in Patients With Drug-resistant Epilepsy
Acronym: IF-MCT16:8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Marburg (Other)
Responsible Party: Principal Investigator, Susanne Knake, Principal investigator, Philipps University Marburg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-92 BO
Record Dates: First submitted 2023-08-08; First posted 2023-08-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy; Intermittent Fasting
Keywords: Drug-resistant epilepsy; Intermittent fasting; Seizure frequency; Biomarkers; Neural networks; Microbiome
MeSH Terms: conditions — Epilepsy; Intermittent Fasting; Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IF 16:8 (Active Comparator): 12 weeks intermittent fasting according to the 16:8 method (IF 16:8)
  Interventions: Other: IF 16:8 as active comparator vs. IF MCT 16:8 as experimental arm
- IF MCT 16:8 (Experimental): 12 weeks intermittent fasting with additional intake of exogenous MCTs (IF MCT 16:8)
  Interventions: Other: IF 16:8 as active comparator vs. IF MCT 16:8 as experimental arm

INTERVENTIONS:
Other: IF 16:8 as active comparator vs. IF MCT 16:8 as experimental arm — 12 weeks intermittent fasting according to the 16:8 method (IF 16:8) are compared with 12 weeks intermittent fasting with additional intake of exogenous MCTs (IF MCT 16:8) in a within-subject-crossover design in 28 patients with drug-resistant epilepsy. In order to enable the highest possible adherence, there are no restrictions on the composition of the food.

SUMMARY:
The objective of the prospective monocentric pilot trial is to investigate the influence of intermittent fasting with or without a once-daily intake with medium chain triglycerides (MCTs) on the frequency of seizures in patients with therapy-refractory epilepsy. The effects of 12 weeks intermittent fasting according to the 16:8 method (IF 16:8) are compared to 12 weeks intermittent fasting with additional intake of exogenous MCTs (IF MCT 16:8) in a within-subject-crossover-design in 28 patients with drug-resistant epilepsy.

DETAILED DESCRIPTION:
One in three patients suffering epilepsy does not become seizure-free with conventional pharmacotherapy. The chance of seizure freedom with each additional medication is only in the single-digit percentage range. For this reason, additive therapies such as the ketogenic diet play an important role. By means of a ketogenic diet, a significant reduction in the frequency of seizures has been shown in various studies for children. The main goal is the body's own production of ketone bodies in the liver, which are used instead of glucose to produce the energy carrier ATP. This metabolic change results in biochemical, metabolic and hormonal changes that may reduce the severity and frequency of epileptic seizures, although the exact mechanisms are not yet understood. Common to all forms of ketogenic diets (e.g. classic kKD, modified Atkins diet, low glycemic index diet) is a specific preparation of each meal with plans for meals and often an initiation of additive therapy in the inpatient setting or by trained staff. Especially in adulthood, the lack of treatment adherence seems to play an important role in the effectiveness of the ketogenic diet. A form of ketogenic diet which might be more suitable for everyday use is intermittent fasting.

The primary aim of the prospective monocentric pilot trial is to investigate the effect of intermittent fasting with and without a once-daily intake of medium-chain triglycerides (MCTs) on the frequency of seizures in patients with therapy-refractory epilepsy. The effects of 12 weeks intermittent fasting according to the 16:8 method (IF 16:8) are compared to 12 weeks intermittent fasting with additional intake of exogenous medium chain triglycerides (IF MCT 16:8) in a within-subject-crossover design in 28 patients with drug-resistant epilepsy. Secondarily, the influence of this diet on the composition of the gut microbiome, the T-cell mediated innate immune system and neuronal signalling pathways and networks will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to provide informed consent
* Drug-resistant epilepsy
* At least 3 seizures per month

Exclusion Criteria:

* Pregnancy
* Breast feeding period
* Metabolic disorder (e.g. diabetes, liver cirrhosis, kidney disease)
* Eating Disorder (e.g. anorexia, bulimia)
* Chronic inflammatory gut disease
* Active cancerous disease
* Antibiotics within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Effect of intermittent fasting according to the 16:8 method with and without exogenous MCTs on seizure frequency in drug-resistant epilepsy | 3 months
  Monthly seizure frequency is recorded using standardized seizure diaries.

SECONDARY OUTCOMES:
Effect of intermittent fasting according to the 16:8 method on therapy adherence in patients with drug-resistant epilepsy | 3 months
  The nutritional behavior during the studio is recorded using a standardized daily nutrition diary.
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on ketosis in patients with drug-resistant epilepsy | 3 months
  All participants measure their ketosis weekly with a standardized ketosis device during the fasting episode and document this in a ketosis table provided.
Effect of intermittent fasting according to the 16:8 method on self-efficacy in patients with drug-resistant epilepsy | 3 months
  Self-efficacy is determined using the scale of general self-efficacy expectation (Jerusalem & Schwarzer). This includes 10 items with 4 degrees. High scores mean a high level of general self-efficacy expectation.
Effect of intermittent fasting according to the 16:8 method on life-quality in patients with drug-resistant epilepsy | 3 months
  Life-quality is measured using the standardized questionnaire on life quality.
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on biomarkers in patients with drug-resistant epilepsy | 3 months
  The metabolome is examined using a mass spectroscopic blood sample. The microbiome is examined using a standardized stool sample using next-generation sequencing.
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on neural networks in patients with drug-resistant epilepsy | 3 months
  Neural networks are measured using magnetic resonance imaging (diffusion tensor imaging and resting state MRI).
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on immune status in patients with drug-resistant epilepsy | 3 months
  The immune status and in particular the T-cell mediated innate immune response is determined serologically.
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on fatigue in patients with drug-resistant epilepsy | 3 months
  Fatigue is measured using the standardized Fatigue-Impact-Scale (FIS)-Test.
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on attention in patients with drug-resistant epilepsy | 3 months
  Attention is measured using the standardized test battery for attention testing (TAP-Test).
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on neurotransmitter gamma-aminobutyric acid (GABA)in patients with drug-resistant epilepsy | 3 months
  The change in the neurotransmitter GABA is examined serologically over the period of the study phase.
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on stress response in patients with drug-resistant epilepsy | 3 months
  Stress response in hair cortisol of all participants is recorded using several hair samples.
Effect of intermittent fasting according to the 16:8 method with exogenous MCTs on intima media thickness in patients with drug-resistant epilepsy | 3 months
  Intima media thickness of all participants will be recorded with a duplex sonographic examination of the arteries supplying the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Wiebke Hahn, MD, Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps University Marburg, Faculty of Medicine, Department of Neurology, Epilepsy Center, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No